CLINICAL TRIAL: NCT00078637
Title: Phase I and Pharmacokinetic Study of E7820 After Oral Administration to Patients With Malignancy
Brief Title: Dosing and Safety Study of E7820 in Patients With a Malignant Solid Tumor or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7820-A001-102
Record Dates: First submitted 2004-03-03; First posted 2004-03-05 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Neoplasms; Lymphoma, Malignant
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — N-(3-cyano-4-methyl-1H-indol-7-yl)-3-cyanobenzene-sulfonamide

INTERVENTIONS:
Drug: E7820

SUMMARY:
This is a first-in-man, open-label, non-randomized, multiple dose, multiple cycle, dose escalation study to determine the MTD, safety, PK, and pharmacodynamics of E7820 in patients with a malignant solid tumor or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed malignant solid tumor or lymphoma. Malignancy must be advanced and require systemic therapy. Malignancy must be one for which no standard therapy is available or the patient must not be a candidate for standard therapy.
* Patients must have a Karnofsky Performance Status of >= 70%,
* Patients must have a life expectancy of >= 3 months,
* Patients must be aged >= 18 years,
* Patients must have adequate renal function as evidenced by serum creatinine <= 1.5 mg/dL or creatinine clearance >= 60 mL/minute/1.73m2,
* Patients must have adequate bone marrow function as evidenced by ANC >= 1,500 mm3 and platelets >= 100,000 mm3, must have adequate liver function as evidenced by bilirubin <= 1.5 mg/dL and alanine transaminase (ALAT) and aspartate transaminase (ASAT) <= 2.5 times the upper limits of normal (ULN) (unless related to liver metastases in which case <= 5 x ULN),
* Patients must be willing and able to comply with the study protocol for the duration of the study, and
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

* Patients who have a history of previous hypersensitivity to sulfonamide derivatives, Patients who have received chemotherapy within 4 weeks (6 weeks if nitrosoureas were received) of commencing study treatment,
* Patients who have had radiation to >= 25% of their bone marrow (e.g., pelvic radiation) within 4 weeks of E7820 treatment,
* Patients who have not recovered from any clinically significant chemotherapy or radiotherapy related toxicity at study entry.
* Patients who have received investigational drugs or other antineoplastic therapy within 28 days of E7820 treatment,
* Patients who have had major surgery within 4 weeks of study drug administration,
* Women who are pregnant or breast-feeding. -- Women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential),
* Fertile men and fertile women who are not willing to use contraception or fertile men or fertile women with a partner who is not willing to use contraception,
* Patients with active central nervous system (CNS) metastases (i.e., evidence of progressive clinical symptoms, edema requiring corticosteroids, or tumors exhibiting growth on sequential MRI or CT scans),
* Patients who are known to be positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus,
* Patients with severe uncontrolled intercurrent illness/infection (excluding malignancies),
* Patients with a history of unstable ischemic disease,
* Patients with a history of clinically significant thrombosis,
* Patients receiving antithrombotic (including aspirin) or therapeutic anticoagulant therapy (prior to study entry, patients receiving these types of drugs must have been off therapy for at least 7 days),
* Patients with a history of documented vascular headache with neurological changes,
* Patients < 30% of ideal weight for height and age according to the Metropolitan Life Insurance Company Statistical Bulletin, or
* Patients with significant disease, or any condition, which in the Investigator's opinion would exclude the patient from the study, or
* Patients who have pulmonary disease that puts them at risk of hemoptysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-01; Primary Completion 2006-08 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jantien Wanders, M.D., Study Director — Eisai Inc.
Locations (1):
- San Antonio, Texas, United States